CLINICAL TRIAL: NCT01159704
Title: Peer Leaders as HIV Risk Reduction Change Agents Among Injection Drug Users (IDUs) in Ukraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 09-0823; R01DA026739-01A1 (NIH)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: HIV Infection; HIV Risk Behaviors
Keywords: HIV infection; Intervention; Risk-reduction; Injection drug users
MeSH Terms: conditions — HIV Infections; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Network plus HIV Counseling&Education (Experimental): Social network peer education model plus HIV testing and counseling; the C & E intervention is a manualized individual-level model consisting of two education and counseling sessions that "structurally bracket confidential HIV antibody screening."
  Interventions: Behavioral: Peer Education Model; Behavioral: HIV Counseling and Education Model
- HIV Counseling and Education (C&E) only (Active Comparator): HIV testing and counseling C&E; the C & E intervention is a manualized individual-level model consisting of two education and counseling sessions that "structurally bracket confidential HIV antibody screening."
  Interventions: Behavioral: HIV Counseling and Education Model

INTERVENTIONS:
Behavioral: Peer Education Model — The peer education intervention will be delivered by trained outreach workers in a group format with 8-10 indexes over five sessions spanning three weeks. The sessions will focus on knowledge of HIV transmission, self-efficacy and skills-building regarding HIV risk reduction, with an emphasis on the dissemination of such information and skills to network members.
  Arms: Network plus HIV Counseling&Education
Behavioral: HIV Counseling and Education Model — The C & E intervention is a manualized individual-level model consisting of two education and counseling sessions that "structurally bracket confidential HIV antibody screening."

SUMMARY:
Using a randomized clinical trial (RCT), this study is designed to assess the effectiveness of HIV (human immunodeficiency virus) risk-reduction interventions targeting injection drug users (IDUs) in three Ukraine oblasts (regions). The investigators propose to compare the effectiveness of a revised and updated manually-driven HIV testing and counseling intervention, the Counseling and Education (C & E) model developed by NIDA, with the C & E plus a manualized network intervention. At each site, Odessa, Donetsk and Nikolayev, 250 "index members" and 500 of their network members will be recruited through street outreach over a 32-month period and randomly assigned to C & E alone or C & E plus the network intervention. Participants will be tested for drug metabolites, interviewed using ACASI (Audio Computer-Assisted Self-Interviewing), and given a rapid test for HIV at baseline, 6 and 12-months. At six-months, network members will be asked to recruit two others they inject with but who are not in the study. Primary outcomes include knowledge, self-efficacy, injection and sex-related risk behavior reduction and partner disclosure among indexes and primary and secondary network members and intervention diffusion to secondary network members. The investigators hypothesize more positive and significant change, including injection and sex risk reduction, intervention diffusion, and partner disclosure, among indexes as well as first and second network members in the network plus C & E arm compared to C & E alone. Specific aims include:

1. To compare the effectiveness of the C & E alone with the additive effect of a network intervention plus C & E in increasing knowledge about HIV and increasing self-efficacy to practice safer injection and sex-related behaviors among indexes, primary and secondary network members.
2. To assess the effectiveness of the C & E alone with the additive effect of a network intervention plus C & E in reducing drug and sex risk behaviors among indexes, primary and secondary network members.
3. To compare the extent of intervention diffusion to second wave network members in the two arms.
4. To evaluate the extent of disclosure by HIV positive indexes and network members in the two arms

ELIGIBILITY:
Inclusion Criteria:

* active drug injector
* 16 years of age or older
* not too intoxicated to give informed consent
* not planning to leave the area in the next 6 months and no pending court date that might result in incarceration
* agree to HIV testing and counseling
* not involved in prior project research activities in teh previous 24 months
* Indexes: must be able to recruit two eligible network members into the study
* Network: agree to participate in five peer educator training sessions

Exclusion Criteria:

* being too intoxicated at the time of the interview
* impaired mentally due to physical or psychological problems to the point that they cannot voluntarily consent to participate in the study and/or respond to the interview
* have a known reason why they will not be available for the intervention or the follow-up interview
* have been involved in prior project research activities in the previous 24 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2304 (Actual)
Dates: Start 2010-07; Primary Completion 2015-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
HIV Knowledge | Follow-up interviews at 6 and 12 months
Self-efficacy regarding HIV risk reduction | Follow-up interviews at 6 and 12 months
Injection risk behavior reduction | Follow-up interviews at 6 and 12 months
Sex-related risk behavior reduction | Follow-up interviews at 6 and 12 months
Intervention diffusion to secondary network members | Follow-up interviews at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Booth, PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- Ukraine (3):
  - NGO, Donetsk
  - NGO, Nikolayev
  - NGO, Odesa

REFERENCES:
- [Derived] Booth RE, Davis JM, Dvoryak S, Brewster JT, Lisovska O, Strathdee SA, Latkin CA. HIV incidence among people who inject drugs (PWIDs) in Ukraine: results from a clustered randomised trial. Lancet HIV. 2016 Oct;3(10):e482-9. doi: 10.1016/S2352-3018(16)30040-6. Epub 2016 Jul 29. PMID 27658879